CLINICAL TRIAL: NCT02246569
Title: Impact of Endoscopic Lung Volume Reduction Via Coils on Inspiratory Muscle Strength in Patients With COPD
Brief Title: Lung Volume Reduction Via Coils in Patients With COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 14-001
Record Dates: First submitted 2014-09-11; First posted 2014-09-22 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic obstructive pulmonary disease (COPD); endoscopic lung volume reduction; RePneu®Coils; physical capacity; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
For patients with emphysema lung volume reduction (ELVR) could be an expedient approach for the reduction of distension of the lung. ELVR may be performed using RePneu® Coils. After the insertion of the coils distended lung sections shrink so that healthy parts can expand.

In the present study investigators intend to examine, whether the insertion of the coils improves diaphragm function and force of the breathing muscles. Investigators hypothesize that reduction of lung volume eliminates or reduces flattening of the diaphragm and relieves breathing muscles, respectively respiratory pump, which aims to reduce dyspnea.

DETAILED DESCRIPTION:
In line with routine explorations it is necessary to clarify whether a patient is suitable for the endoscopic lung volume reduction. To address this question lung function diagnostics, 6-minutes-walk-test, blood withdrawal, CT of the thorax, lung perfusion scintigraphy and transthoracic echocardiography have to be performed.

After confirmation of the suitability for the endoscopic lung volume reduction patients who fulfill all other eligibility criteria will be educated about the aim and performance of the study by an investigator. After reading the patient information patient may submit his informed written consent. After that information on the risks will be given by a treating physician.

Following examination will be performed additional due to the study: determination of the strength of breathing muscles, determination of the life quality index via St.-George-questionary and determination of the depression score via SF-8-questionary (short form-8).

After that coils will be implanted and a permanent post-operative examination will be performed for 24 hours.

Three, respectively nine month after the implanting follow up exploration will be performed on the study patients.

ELIGIBILITY:
Inclusion Criteria:

* bilateral lung emphysema after CT with sufficient amount of tissue to perform RePneu Coil implantation at the discretion of the treating physicians
* homogeneous or heterogeneous emphysema
* previous guidelines-based therapy of COPD (including vaccinations against Pneumococcal infections and seasonal influenza)
* nicotine abstention for not less than three months, documented by CO-HB (haemoglobin) < 2%
* FEV 1 (Forced Expiratory Volume 1 / one second capacity) ≤ 45% of reference value, after bronchodilatation
* total lung capacity (TLC) ≥ 100% of reference value
* residual volume (RV) ≥ 175% of reference value
* patient's suitability for endoscopic lung volume reduction according to multidisciplinary decision of pneumology and thorax surgery division.
* signed Informed Consent
* understanding of the nature, significance and implications of the study
* ability to understand and follow instructions of the study stuff

Exclusion Criteria:

* echo-cardiographic right ventricular pressure (PAPsys) > 50 mmHg
* indication for a permanent anticoagulation therapy (besides ASS)
* pulmonal cachexia
* pregnancy and lactating
* permanent treatment with > 20 mg Prednison per day
* hospitalisation due to a COPD-exacerbation in the last 3 months
* > 3 steroid-treated exacerbations in the last year
* Increase of FEV1 (Forced Expiratory Volume) ≥ 20% after bronchodilatation
* severe diffusion impairment (DLCO < 20%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with severe COPD (GOLD stage III or IV)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
breathing strength | Change of breathing strength 3 (respectively 9) months after the bronchoscopy
  Maximal Inspiratory Pressure (PImax) Maximal Expiratory Pressure (PEmax) Neuromuscular drive (P0.1) Sniff nasal pressure

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dreher, Univ.-Prof., Principal Investigator — RWTH University Hospital MK1
Locations (1):
- RWTH Univerity Hospital MK1, Aachen, Germany